CLINICAL TRIAL: NCT06969300
Title: Efficacy and Safety Evaluation of Fractional Microneedling Radiofrequency Combined With 30% Supramolecular Salicylic Acid in the Treatment of Refractory Erythrotelangiectatic Rosacea
Brief Title: FMRF Combined With 30% SSA in the Treatment of Rosacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Weihui Zeng, professor, Second Affiliated Hospital of Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MR-61-24-008032
Record Dates: First submitted 2025-04-29; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Rosacea
Keywords: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Salicylic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gold micro-needling treatment (Other): The treatment (with gold microneedles) was administered on the day of enrollment after the completion of the detection items. Follow-up visits were conducted at 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks. The follow-up contents included visia photography, camera photography, non-invasive skin examination, questionnaire assessment, etc. The study duration was 12 weeks.
  Interventions: Device: Gold micro needles
- Gold micro-needling combined with salicylic acid treatment (Experimental): On the day of enrollment, the treatment was carried out after the completion of the detection items (gold microneedle + 30% salicylic acid on half of the face). A site follow-up was conducted one week later, and then follow-ups were conducted every two weeks for the second and third acid brushing treatments. Follow-up visits were also conducted every four weeks at the 8th and 12th weeks. The follow-up contents included: Visia photography, camera photography, non-invasive skin examination, questionnaire assessment, etc. The study duration was 12 weeks.
  Interventions: Drug: Gold micro-needles combined with salicylic acid

INTERVENTIONS:
Device: Gold micro needles — The treatment (with gold microneedles) was administered on the day of enrollment after the completion of the detection items. Follow-up visits were conducted at 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks. The follow-up contents included visia photography, camera photography, non-invasive skin examination, questionnaire assessment, etc. The study duration was 12 weeks.
  Arms: Gold micro-needling treatment
Drug: Gold micro-needles combined with salicylic acid — On the day of enrollment, the treatment was administered (gold microneedle + 30% salicylic acid on half of the face) after the completion of the detection items. A site follow-up was conducted one week later, and a follow-up was carried out two weeks later with the second acid brushing treatment. A follow-up was conducted four weeks later with the third acid brushing treatment. Follow-up was also conducted at the eighth and twelfth weeks. The follow-up contents included: Visia photography, camera photography, non-invasive skin examination, questionnaire assessment, etc. The study duration was 12 weeks.
  Arms: Gold micro-needling combined with salicylic acid treatment

SUMMARY:
This study was a single-center, case-by-case, bilateral facial comparison study. A total of 15 patients were included. On the day of enrollment, after the completion of the test items, treatment was carried out (full face gold micro-needling + 30% salicylic acid on the half face), and on-site follow-up was conducted 1 week later, 2 weeks later follow-up was conducted and the second acid brushing treatment was performed, 4 weeks later follow-up was conducted and the third acid brushing treatment was performed, on-site follow-up was conducted at the 8th week and the 12th week, and the follow-up contents included: Visia photography, camera photography, non-invasive skin testing, questionnaire assessment, etc. The study duration was 12 weeks.

DETAILED DESCRIPTION:
This study is a single-center case-control study with half-side face as the control group. According to the inclusion and exclusion criteria, 15 patients with rosacea (erythema and telangiectasia type) were included. Before and after treatment, various skin indicators of the patients were evaluated and followed up. Through screening, subjects who met all the inclusion criteria and did not violate any of the exclusion criteria would be included in this study. The researchers measured and evaluated the various skin indicators of the patients. On the day of enrollment, the project was completed and treatment was carried out (full face gold micro-needling + 30% salicylic acid on half-side face), and then on-site follow-up was conducted 1 week later, 2 weeks later, 4 weeks later, 8 weeks later, and 12 weeks later. The follow-up contents included: Visia photography, camera photography, non-invasive skin detection, questionnaire assessment, etc. The study duration was 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. According to the latest diagnostic criteria of the American Rosacea Society (2017 version) - Annex 1, patients diagnosed with the main phenotype of erythema and telangiectasia.
2. The therapeutic response to the medication is unsatisfactory and the condition is prone to relapse.
3. Age range: 18 to 60 years old
4. The patient voluntarily participated in this clinical study and signed the written informed consent form.

Exclusion Criteria:

1. The patient has other skin disorders on the face, such as melasma, freckles and seborrheic dermatitis, which may affect the judgment of the test results.
2. Individuals who are allergic to the test drug or have hypersensitive constitution.
3. Patients who are pregnant, about to become pregnant or are lactating.
4. Patients with acne during the consultation.
5. Patients who had undergone facial injections or surgeries within the past two months before the trial.
6. Patients with immunodeficiency diseases and abnormal coagulation function.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
The range, quantity and degree of facial erythema | Before the first treatment, 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks
  After cleansing the face with Visia, take a rest for 30 minutes at room temperature of 25 degrees Celsius and then take frontal and lateral images.
Erythema score | Before the first treatment, 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks
  Assessment of lesion morphology score: No visible erythema under natural light = 0 points; Mild erythema can be observed under natural light, presenting as pale red, not obvious at a distance of 50 cm, and can be covered by simple makeup or beard covering = 2 points; Moderate erythema can be observed under natural light, presenting as red, obvious at a distance of 50 cm, and simple makeup or beard covering is not sufficient to cover = 4 points; Severe erythema can be observed under natural light, presenting as bright red, still obvious at a distance of more than 50 cm, and simple makeup or beard covering is insufficient to cover = 6 points. Weighted coefficient for the number/area of lesions: 1-10/5%-10% = 1, 11-20/11%-20% = 2, >20/20% = 3. Total score of lesion severity = Morphology score × Weighted coefficient. Based on the score, calculate the therapeutic index, therapeutic index = (Total score before treatment - Total score after treatment) / Total score before treatment × 100%
TEWL | Before the first treatment, 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks
  The skin non-invasive detector conducts the test.
MI | Before the first treatment, 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks
  The skin non-invasive detector conducts the test.
L*a*b | Before the first treatment, 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks
  The skin non-invasive detector conducts the test.
The moisture content of the stratum corneum | Before the first treatment, 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks
  The skin non-invasive detector conducts the test.
Skin elasticity | Before the first treatment, 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks
  The skin non-invasive detector conducts the test.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No